CLINICAL TRIAL: NCT01253005
Title: The Effect of Physical Properties of Lipid Emulsions on Gastrointestinal Motility and Transit, Hormonal Feedback, Visceral Sensation and Satiety in Healthy Volunteers
Brief Title: The Effect of Physical Properties of Lipid Emulsions on Gastrointestinal Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: SNF 320030_0-0197
Record Dates: First submitted 2010-09-29; First posted 2010-12-03 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Healthy Controls

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Behavioral: Nutritional intervention — This study will investigate the effects of particle size of different triglyceride emulsions as well as the dynamics of intragastric structure formation and breakdown of the emulsions on GI function, the kinetics of the endocrine and the satiation response in healthy volunteers.

SUMMARY:
This study will investigate the effects of particle size of different triglyceride emulsions as well as the dynamics of intragastric structure formation and breakdown of the emulsions on GI function, the kinetics of the endocrine and the satiation response in healthy volunteers. 12 healthy participants will be studied on four occasions on four separate days in a double blind randomized design

DETAILED DESCRIPTION:
The mechanisms by which food structure impacts on lipid digestion and the subsequent metabolic processes, including the impact on satiety and satiation, are relatively unexplored, but may have great consequences on the development of effective strategies for weight management. Data from previous studies suggest that (i) the droplet size of a fat emulsion has a distinct influence on GI function and visceral perception (ii) that the biomechanical and digestive properties of the human gut may induce micro structural changes to specifically designed lipid emulsions resulting in different patterns of lipolysis.

The study will assess the effects of triglyceride emulsion with different particle (0.6, 30 μm) sizes and sensitivities to the acidic and shear environment of the stomach on GI function and the kinetics of endocrine and satiation response.

In this study healthy participants will be studied on four occasions on four separate days in a double blind randomized design. The assessment of gastric function will be monitored by novel MRI techniques and breath tests and neurohormonal response by blood sampling.

ELIGIBILITY:
Inclusion criteria:

* Body mass index (BMI): 18.5-24.9 kg/m2,
* Able to communicate well with the investigators
* Provide written consent

Exclusion criteria:

General exclusion criteria:

* Psychiatric (DSM IV) disorders limiting the ability to comply with study requirements
* Epilepsy
* Presence of metallic implants, devices or metallic foreign bodies
* Use of medications influencing upper GI motility within one week of the study (i.e. calcium channel blockers, prokinetic drugs, macrolide antibiotics)
* Evidence of current drug or alcohol abuse
* Previous history of gastrointestinal disease or surgery of the upper GI tract except appendicectomy or hernia repair
* Pregnancy and lactation period

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The GI response to lipid emulsions with different particle sizes and sensitivities to the acidic and shear environment of the stomach in terms of: motility, neurohormonal feedback, sensation and satiety | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fried, Professor MD, Principal Investigator — University Hospital Zurich, Gastroenterology and Hepatology
Locations (1):
- University Hospital Zurich, Gastroenterology and Hepatology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Steingoetter A, Buetikofer S, Curcic J, Menne D, Rehfeld JF, Fried M, Schwizer W, Wooster TJ. The Dynamics of Gastric Emptying and Self-Reported Feelings of Satiation Are Better Predictors Than Gastrointestinal Hormones of the Effects of Lipid Emulsion Structure on Fat Digestion in Healthy Adults-A Bayesian Inference Approach. J Nutr. 2017 Apr;147(4):706-714. doi: 10.3945/jn.116.237800. Epub 2017 Feb 22. PMID 28228504
- [Derived] Steingoetter A, Radovic T, Buetikofer S, Curcic J, Menne D, Fried M, Schwizer W, Wooster TJ. Imaging gastric structuring of lipid emulsions and its effect on gastrointestinal function: a randomized trial in healthy subjects. Am J Clin Nutr. 2015 Apr;101(4):714-24. doi: 10.3945/ajcn.114.100263. Epub 2015 Feb 25. PMID 25833970